CLINICAL TRIAL: NCT05490706
Title: The Influence of Different At-home Exercise Strategies on 24h Glycemic Control in Women at Risk for With Metabolic Disease
Brief Title: The Influence of Different At-home Exercise Strategies on 24h Glycemic Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Responsible Party: Principal Investigator, Jenna Gillen, Assistant Professor, University of Toronto
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 42756-2
Record Dates: First submitted 2022-07-29; First posted 2022-08-08 (Actual); Last update posted 2023-05-15 (Actual); Status verified 2023-05

CONDITIONS: Metabolic Disturbance
Keywords: women; glycemic control; exercise
MeSH Terms: conditions — Motor Activity | interventions — Walking

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Bodyweight interval exercise (Experimental): Performing 15 minutes of bodyweight interval exercise after dinner
  Interventions: Behavioral: Bodyweight interval exercise
- Walking (Experimental): Performing a 30 minute walk after dinner
  Interventions: Behavioral: Walking
- Non exercise control (No Intervention): Performing no exercise after dinner

INTERVENTIONS:
Behavioral: Bodyweight interval exercise — Performing 15 minutes of bodyweight interval exercise after dinner at home by following a video
  Arms: Bodyweight interval exercise
Behavioral: Walking — Performing a 30 minute minute walk after dinner at home
  Arms: Walking

SUMMARY:
This study will determine how different at-home exercise strategies influence 24hr glycemic control in women with metabolic dysfunction.

DETAILED DESCRIPTION:
Elevations in blood glucose concentration increase risk for cardiometabolic diseases including type 2 diabetes and cardiovascular diseases. Exercise can improve glycemic control, but there is limited research comparing the effectiveness of different exercise strategies in women. The aim of this study is to examine, under free-living conditions, how performing either walking and bodyweight interval exercise after dinner influences glycemic control in women with or at risk for type 2 diabetes. Glycemic control will be measured with continuous glucose monitors.

ELIGIBILITY:
Inclusion Criteria:

* Females
* no cancer history
* ≥50 years old
* Have metabolic dysfunction (defined as self-reported diagnosis of pre-diabetes, type 2 diabetes, or at least moderate Canadian diabetes risk (CANRISK) score)
* Owns a smartphone with Bluetooth capability with Apple or Android operating system
* deemed safe to exercise as per the CSEP Get Active Questionnaire
* Enrolled in NCT05454943

Exclusion Criteria:

* Type 1 diabetes
* Taking exogenous insulin, sulfonylureas, or GLP-1 receptor agonists
* Self-reported history of an eating disorder
* BMI <18.5 kg/m
* Working night or rotating shifts
* Eating window <12 hours or consistently eating less than 3 meals/day in the past 3 months
* Major dietary changes within the past 3 months (i.e. calorie counting, ketogenic diet)

Min Age: 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2022-07-07 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
24hr Glucose area under the curve | 24 hours
  Glucose area under the curve over 24hr

SECONDARY OUTCOMES:
24hr Average glucose concentration | 24 hours
  Average glucose concentration over 24 hr
Postprandial dinner glucose response | 2 hours
  Measured as the 2hr postprandial glucose incremental area under the curve (iAUC), average glucose and peak glucose
Postprandial breakfast glucose response | 2 hours
  Measured as the 2hr postprandial iAUC, average glucose and peak glucose
Postprandial lunch glucose response | 2 hours
  Measured as the 2hr postprandial glucose iAUC, average glucose and peak glucose
Nocturnal glucose | ~6-8 hours
  Measured as the overnight glucose average and AUC
Time in hyperglycemia | 24 hours
  Time (minutes and percent per day) above 10mmol/L over 24hr
Time in hypoglycemia | 24 hours
  Time (minutes and percent per day) under 3.9mmol/L over 24 hr
Time in range | 24 hours
  Time (minutes and percent per day) above 3.9 but under 10mmol/L
Continuous overall net glycemic action (CONGA) | 24 hours
  Calculated measure of glycemic variability
Change in glucose during exercise | 15-30 minutes
  Post vs. pre glucose concentration around exercise
Mean amplitude glycemic excursion (MAGE) | 24 hours
  Calculated measure of glycemic variability
Standard deviation (SD) | 24 hours
  Calculated measure of glycemic variability
% coefficient of variation (CV) | 24 hours
  Calculated measure of glycemic variability

CONTACTS AND LOCATIONS:
Overall Officials: Jenna Gillen, PhD, Principal Investigator — University of Toronto
Locations (1):
- University of Toronto, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No